CLINICAL TRIAL: NCT02885480
Title: ROUTE PATIENT CONSULTANT in OUTPATIENT CARE PSYCHIATRIC EMERGENCY SERVICES AND PUBLIC OF EUROMETROPOLE STRASBOURG
Brief Title: Courses Emergency Psychiatric Strasbourg
Acronym: PUPS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 5884
Record Dates: First submitted 2016-08-26; First posted 2016-08-31 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-09

CONDITIONS: Psychiatric Emergency
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: questionnaires

SUMMARY:
Describe and analyze routes and modes of care for patients in emergency consultant in various emergency care and public psychiatric outpatient devices to provide useful information to optimize trajectories taken into psychiatric load on the Eurométropole territory upstream and downstream of where they viewed urgently.

ELIGIBILITY:
Inclusion Criteria:

* All patients, men and women, adults and minors of 11 years and more, seen for psychiatric consultation request emergency (unscheduled and requiring specialized psychiatric consultation within 72 hours)

Exclusion Criteria:

* Will not be included in the study psychiatric consultations requested by internal hospital services other than emergency services, patients with psychiatric emergencies revised for post-emergency consultations

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients treated in psychiatric emergencies
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
management of emergency patients consulting | follow-up of 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Pierre VIDAILHET, MD, Principal Investigator — Les Hôpitaux Universitaires de Strasbourg
Locations (1):
- Les Hôpitaux Universitaires, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No